CLINICAL TRIAL: NCT03521856
Title: Trial for Shoulder Pathology and Pain in Chronic SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Roy Felix, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20111005
Record Dates: First submitted 2018-04-29; First posted 2018-05-11 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Shoulder Pain
Keywords: spinal cord injuries; SCI
MeSH Terms: conditions — Shoulder Pain; Spinal Cord Injuries | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shoulder exercise intervention (Experimental): A home exercise intervention for strengthening and stretching the shoulders - Strengthening and Optimal Movement for Painful Shoulders (STOMPS) - performed 3 times per week for 12 weeks.
  Interventions: Behavioral: shoulder exercise
- education-only control (Active Comparator): Subjects watched a 1 hour educational video on shoulder anatomy, mechanisms of shoulder injury and pain, and hints for managing shoulder pain
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: shoulder exercise — Exercises performed 3 times a week for 12 weeks
  Arms: shoulder exercise intervention
Behavioral: education
  Arms: education-only control

SUMMARY:
This research study will investigate in a 12-week home exercise program to see whether it is effective in improving shoulder pathology and reducing shoulder pain in persons with chronic spinal cord injury. The research study will involve ultrasound shoulder examinations of your shoulders using a non-invasive medical ultrasound machine, as well as clinical shoulder examinations and completion of a number of pain questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Candidates will be men or women, 18 years of age or older.
2. Candidates must have an SCI and be at least 1 year post-diagnosis
3. Candidates must use a wheelchair (manual or electric) for at least the majority of the time.
4. Candidates must be able to transfer themselves without the help of others.
5. The presence of at least moderate shoulder pain (rating of >= 4 on a 0-10 rating scale for average pain intensity) for 3 or more months.

Exclusion Criteria:

1. Patients younger than 18 years of age.
2. Patients who have a history of pre-injury rotator cuff tears or shoulder injury.
3. Patients who do not use a wheelchair (manual or electric) at least 50% of the time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Change in shoulder pathology | Baseline to week 12
  Quantitative ultrasound measures of the supraspinatus tendon

SECONDARY OUTCOMES:
Change in shoulder pain using the numerical rating scale | Baseline to week 12
  Numerical rating scale for pain intensity (0 = no pain; 10 = most intense pain imaginable)
Change in shoulder pain using the numerical rating scale | Baseline to week 16
  Numerical rating scale for pain intensity (0 = no pain; 10 = most intense pain imaginable)
Change in shoulder pain using the WUSPI | Baseline to week 12
  Wheelchair Users Shoulder Pain Index (WUSPI) (0 - 150)
Change in shoulder pain using the WUSPI | Baseline to week 16
  Wheelchair Users Shoulder Pain Index (WUSPI) (0 - 150)
Change in shoulder pathology | Baseline to week 16
  Quantitative ultrasound measures of the supraspinatus tendon

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Felix, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulroy SJ, Thompson L, Kemp B, Hatchett PP, Newsam CJ, Lupold DG, Haubert LL, Eberly V, Ge TT, Azen SP, Winstein CJ, Gordon J; Physical Therapy Clinical Research Network (PTClinResNet). Strengthening and optimal movements for painful shoulders (STOMPS) in chronic spinal cord injury: a randomized controlled trial. Phys Ther. 2011 Mar;91(3):305-24. doi: 10.2522/ptj.20100182. Epub 2011 Feb 3. PMID 21292803
- [Result] Cardenas DD, Felix ER, Cowan R, Orell MF, Irwin R. Effects of Home Exercises on Shoulder Pain and Pathology in Chronic Spinal Cord Injury: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2020 Jun;99(6):504-513. doi: 10.1097/PHM.0000000000001362. PMID 31851011